CLINICAL TRIAL: NCT05753839
Title: The Role of Cytoreductive Nephrectomy in Metastatic Renal Cell Carcinoma in Immuno-oncology Era: SEVURO-CN Trial
Acronym: SEVURO-CN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1453
Record Dates: First submitted 2023-01-17; First posted 2023-03-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Kidney Cancer; Clear Cell Renal Cell Carcinoma Metastatic; Synchronous Neoplasm
MeSH Terms: conditions — Kidney Neoplasms; Clear-cell metastatic renal cell carcinoma; Neoplasms, Multiple Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upfront cytoreductive nephrectomy (Experimental): Cytoreductive nephrectomy±metastasectomy, followed by induction therapy with nivolumab plus ipilimumab combination and maintenance therapy with nivolumab.
  Interventions: Procedure: Cytoreductive nephrectomy±metastasectomy
- Deferred cytoreductive nephrectomy (Experimental): Cytoreductive nephrectomy±metastasectomy after induction therapy with nivolumab plus ipilimumab combination, followed by maintenance therapy with nivolumab.
  Interventions: Procedure: Cytoreductive nephrectomy±metastasectomy
- No surgery (Active Comparator): Induction therapy with nivolumab plus ipilimumab combination, followed by maintenance therapy with nivolumab.
  Interventions: Other: Human-derived materials sampling

INTERVENTIONS:
Procedure: Cytoreductive nephrectomy±metastasectomy — Partial or complete nephrectomy by open, laparoscopic, or robotic approach and/or metastasectomy Tumor tissue, blood, urine and stool specimens for translational biomarker research will be sample at baseline, surgery, after induction therapy, and after 3 months of maintenance therapy.
  Other Names: Human-derived materials sampling
  Arms: Upfront cytoreductive nephrectomy
Procedure: Cytoreductive nephrectomy±metastasectomy — Partial or complete nephrectomy by open, laparoscopic, or robotic approach and/or metastasectomy Tumor tissue, blood, urine and stool specimens for translational biomarker research will be sample at baseline, surgery, after induction therapy, and after 3 months of maintenance therapy.
  Other Names: Human-derived materials sampling
  Arms: Deferred cytoreductive nephrectomy
Other: Human-derived materials sampling — Tumor tissue, blood, urine and stool specimens for translational biomarker research will be sample at baseline, after induction therapy, and after 3 months of maintenance therapy.
  Arms: No surgery

SUMMARY:
BACKGROUND: The role of cytoreductive nephrectomy (CN) in the treatment of metastatic renal cell carcinoma (mRCC) has been questioned and remains undetermined in the immuno-oncology era. Results from the two randomized trials, CARMENA and SURTIME, have questioned the role and timing of the surgery in these patients, however, these trials have only used the targeted therapy, sunitinib. With the advent of more effective systemic therapies including immune checkpoint inhibitors (ICIs), the role of surgical therapy should be reexamined.

RATIONALE: The therapeutic effects of ICIs have demonstrated improved oncological outcomes compared to sunitinib. The updated results reported the beneficial role of upfront and deferred CN approach for selected patients. No studies have formally investigated the role of CN in the immune-oncology era where combinatorial use of CN plus ICIs might be beneficial.

HYPOTHESIS: Upfront or deferred CN will improve oncological outcomes (overall survival, and progression free survival) in patients with synchronous mRCC and ≤3 IMDC risk features compared to immune checkpoint inhibitors (nivolumab plus ipilimumab combination) alone.

This is an open, randomized, multicenter comparison trial, designed to evaluate the effect of the potential role of CN in combination with immunotherapy in mRCC patients with IMDC intermediate and poor risk.

ELIGIBILITY:
Inclusion Criteria:

1. Core needle biopsy proven metastatic renal cell carcinoma - clear cell histologic subtypes only acceptable.
2. Synchronous metastatic renal cell carcinoma with the primary tumor present in the kidney.
3. Patient must be willing to provide their human-derived materials.
4. Age ≥19.
5. Signed written informed consent obtained prior to any study specific procedures.
6. Patient must be willing and able to comply with the protocol.
7. Measurable disease as per RECIST v 1.1
8. Life expectancy of greater than 4 months.
9. Patients with more than one prognostic factor by the International Metastatic RCC Database Consortium (IMDC) criteria (intermediate- or poor-risk group).
10. Patients for which Nivolumab/Ipilimumab considered indicated according to the recommendations by the national health authorities. The prescription of nivolumab/ipilimumab in the circumstances of the study is considered as a standard treatment.
11. Karnofsky Performance status ≥70
12. Females with a negative serum pregnancy test unless childbearing potential can be otherwise excluded (postmenopausal, hysterectomy or oophorectomy) and not lactating.
13. Fertile women of childbearing potential (<2 years after last menstruation) and men must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgical sterilization).
14. The required laboratory values are as follows:

    * Adequate bone marrow function (Absolute neutrophil count > 1500/mm3, platelets > 100 x 103/µl, hemoglobin > 10.0 g/dL.)
    * International normalized ratio (INR) ≤ 1.2 x upper limit of normal (ULN)
    * Adequate hepatic function (bilirubin ≤ 1.5 x ULN, ALAT ≤ 2.5 x ULN)
    * Adequate kidney function (eGFR > 35 mL/min)

Exclusion Criteria:

1. Prior systemic treatment for mRCC
2. Major surgical procedure, open surgical biopsy, or significant traumatic injury within 28 days prior to enrollment
3. Other cancer within 5 years.
4. Clinically significant (i.e active) cardiovascular disease for example cerebrovascular accidents (< 6 months before inclusion), myocardial infarction (< 6 months before inclusion), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure.
5. No symptomatic brain metastasis requiring systemic corticosteroids (> 10 mg daily prednisone equivalent)
6. Recent (within the 30 days prior to inclusion) treatment with another investigational drug or participation in another investigational study.
7. Any active or recent history of a known or suspected autoimmune disease or recent history of a condition that require systemic corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications, excluding inhaled steroids and topical steroids. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, psoriasis not requiring systemic treatment are permitted to enroll.
8. Oral or i.v. antibiotics administered 14 days prior to initiation of systemic therapy.
9. Any positive test for hepatitis B- or C-Virus indicating acute or chronic infection.
10. Known hypersensitivity to monoclonal antibodies.
11. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
12. Patients disagreeing to provide their human-derived materials.
13. Patients not willing and able to comply with the protocol.
14. Vulnerable subjects (such as children, prisoners, pregnant women, mentally disabled persons, or economically or educationally disadvantaged persons).
15. Patients who cannot read and understand the consent form. (illiterate, foreigners, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2027-12-27 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years follow-up
  Calculated from the date of inclusion, to the date of death of any cause or censored at the date at last follow-up.

SECONDARY OUTCOMES:
Progression free survival | 5 years follow-up
  According to the RECIST v1.1
Objective response rate | 5 years follow-up
  According to the RECIST v1.1
Number of participants with treatment-related adverse events | 5 years follow-up
  By Common Terminology Criteria for Adverse Events version 5.0
Number of participant with surgical morbidity assessed according to the Clavien-Dindo classification of surgical complications | 5 years follow-up
  Assessed according to the Clavien-Dindo classification of surgical complications
Tumor infiltrating lymphocytes | 5 years follow-up
  Measured by flowcytometry at baseline and after surgery and/or after ICIs compared with OS, PFS, ORR
Genetic mutation profiles of primary tissue | 5 years follow-up
  Measured by Next generation sequencing (NGS) methods compared with OS, PFS, and ORR
Genetic mutation profile of circulating tumor DNA | 5 years follow-up
  Measured by NGS methods compared with OS, PFS, and ORR
Genetic mutation profile or urine tumor DNA | 5 years follow-up
  Measured by NGS methods compared with OS, PFS, and ORR
Profile of gut microbiome | 5 years follow-up
  Evaluate the microbiome composition measured by NGS methods compared with OS, PFS, and ORR
Profile of urine microbiome | 5 years follow-up
  Evaluate the microbiome composition measured by NGS methods compared with OS, PFS, and ORR

CONTACTS AND LOCATIONS:
Overall Officials: Won Sik Ham, Principal Investigator — Department of Urology and Urological Science Institute, Yonsei University College of Medicine
Locations (3):
- South Korea (3):
  - Gangnam Severance Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Yongin Severance Hospital, Yongin-si

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JS, Kim J, Jeon J, Lee J, Jang WS, Lee SH, Han WK, Choi YD, Koo KC, Cho KS, Chung BH, Ham WS. The role of cytoreductive nephrectomy in metastatic renal cell carcinoma in immune-oncology era (SEVURO-CN): study protocol for a multi-center, prospective, randomized trial. Trials. 2024 Jul 3;25(1):447. doi: 10.1186/s13063-024-08234-2. PMID 38961439